CLINICAL TRIAL: NCT02274220
Title: Randomized Study of Early Nutritional Delivery on Glucose Control, Insulin Resistance and Systemic Inflammation Following Pediatric Cardiac Surgery
Brief Title: Feeding Study - Effects Post-cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Alejandro Floh, Dr., The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1000046036
Record Dates: First submitted 2014-10-20; First posted 2014-10-24 (Estimated); Last update posted 2018-05-25 (Actual); Status verified 2018-05

CONDITIONS: Heart Disease; Dietary Modification; Insulin Resistance
Keywords: systemic inflammation; glucose metabolism; glucose-insulin ratio
MeSH Terms: conditions — Heart Diseases; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Rapid Advancement of Feeds (Experimental): Postoperative feeds are initiated on first postoperative day and rapidly advanced over 27 hours.
  Interventions: Dietary Supplement: Rapid advancement of feeds
- Average feeding protocol (Experimental): Postoperative feeds are initiated on first postoperative day and advanced in using a standardized protocol that best-reflects current feeding practice. Maximum feeding volume is reached at 60 hours.
  Interventions: Dietary Supplement: Standard advancement of feeds
- Feeds not affected (No Intervention): Postoperative feeds for patients not eligible for randomization are initiated by the treating clinical team and increased as per clinical team's preference.

INTERVENTIONS:
Dietary Supplement: Rapid advancement of feeds — Feeding is initiated on first postoperative day. Bolus feeds are started at 1 mL/kg every three hours and up-titrated by 1 mL/kg every feed (Q 3 hours) to a goal of 10 mL/kg/feed (equivalent to approximately 50 kcal/kg/day). Feeding volume will exceed 20 mL/kg/day by 6 hours following protocol initiation and reach target feeds by 27 hours of protocol initiation.
  Arms: Rapid Advancement of Feeds
Dietary Supplement: Standard advancement of feeds — Feeding is initiated on first postoperative day. Bolus feeds are started at 3 mL every three hours for 24 hours. Bolus feeds then up-titrated by 1 mL/kg every-other feed (Q 6 hours) for 24 hours. Bolus feeds then up-titrated by 1mL/kg every feed for to a goal of 10 mL/kg/feed (equivalent to approximately 50 kcal/kg/day). Feeding volume will reach target feeds by 60-63 hours after protocol initiation.
  Arms: Average feeding protocol

SUMMARY:
The purpose of this randomized trial is to clarify the role of enteral nutrition (EN) on the relationship between cardiopulmonary bypass-induced inflammation and insulin resistance by investigating the effects of two different feeding strategies in infants following cardiac surgery. The study's primary objective is to determine if early and higher volume feeding modifies the relationship between the severity of postoperative systemic inflammation and insulin resistance.

DETAILED DESCRIPTION:
Good nutrition is important for patients after surgery. Patients who are given food tend to have fewer infections, better wound healing, and are possibly discharged more quickly from the intensive care unit and hospital. However, the best time to start feeds and the speed at which they can be increased is unclear. This may be particularly true for young children who have undergone heart surgery using a heart-lung bypass machine (bypass surgery). Bypass surgery can cause inflammation that can change the way the body uses energy and nutrients. Specifically, after bypass the body can become insensitive to insulin (insulin resistant), which means that the cells in the body don't take up sugar from the blood like they are supposed to, and this may lead to complications from the surgery. In a recent study we found that inflammation and insulin resistance was not associated with as many complications in children who were being fed. We are not sure if feeding changed the way in which the body responded after surgery or if doctors chose to feed only patients who were already recovering well. In general, doctors often hesitate to feed patients immediately after surgery because they worry that the body may not be ready for food although there is not much information to prove that this worry is correct. Starting feeds early using a structured feeding plan may be good during the recovery from heart surgery, even in our most vulnerable patients. We therefore designed this study to see if starting feeds early after bypass surgery and increasing them more quickly than our usual routine would decrease inflammation and insulin resistance. We will only study children younger than 6 months of age because they are at higher risk of complications from bypass surgery.

ELIGIBILITY:
Inclusion Criteria:

* less than 6 months of age
* weight > 2.5kg
* surgery using cardiopulmonary bypass
* expected duration of ventilation > 6 hours

Exclusion Criteria:

* cardiac transplantation
* prematurity (<37 weeks gestation AND under 28 days of life)
* intrauterine growth restriction
* NEC
* structural gastrointestinal anomalies
* known preoperative feeding intolerance
* diabetes or known metabolic disorder
* preoperative liver or renal dysfunction
* postoperative contraindication to enteral feeding as determined by clinical team
* previous enrollment at an earlier operation
* in the opinion of the clinical or research team the patient is too well to participate, such that slow escalation to feeds would lead to hunger and therefore be considered inappropriate.

Ages: 1 Minute to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 86 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Insulin resistance | 96 hours
  Plasma insulin concentrations and glucose-insulin ratio (GIR) - GIR will be calculated at each time point and used to reflect insulin resistance, with lower values representing increased resistance

SECONDARY OUTCOMES:
Postoperative systemic inflammation | 96 hours
  Serial measurements of postoperative cytokine (IL-1beta, IL-6, IL-8, IL-10 and TNFalpha) concentrations
Cardiac output | 96 hours
  Postoperative cardiac output measured by respiratory mass spectrometry and Fick equation
Morbidity score | 96 hours
  Postoperative morbidity assessed by a composite morbidity score that includes death, cardiac arrest, use of extracorporeal membrane oxygenation, cardiogenic shock, acute kidney injury, hepatic injury, or hospital-acquired infection.
Number of subjects achieving goal feeds | 96 hours
Number of subjects with NEC/feeding intolerance/protocol violations | 96 hours

CONTACTS AND LOCATIONS:
Overall Officials: Steve Schwartz, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No